CLINICAL TRIAL: NCT00683956
Title: Evaluation of a Closed-Loop Control System for Patient-Specific Induction and Maintenance of Propofol Hypnosis
Brief Title: Evaluation of a Closed-Loop Control System for Administering Patient-Specific Anesthesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: SU-05062008-1141; 13305
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Propofol

INTERVENTIONS:
Device: ReinLoop control software for patient-specific induction and maintenance of anesthesia
Drug: Propofol

SUMMARY:
Numerous efforts have focused on the development of closed-loop systems to control anesthesia using the electrical activity of the brain (EEG) and EEG-based parameters as surrogate measures of anesthetic depth. New systems have been recently developed to considerably improve anesthetic control using model-based, patient-adaptive methods. The purpose of this study is to evaluate the clinical efficacy of a new intelligent software, ReinLoop, in delivering closed-loop, patient-specific hypnosis.

ELIGIBILITY:
Inclusion Criteria:

1. 18-45 years of age
2. Body mass index (BMI) lower or equal to 25 m2/kg
3. Subjects must be able to comprehend spoken and written English

Exclusion Criteria:

1. Any type of psychiatric, neurological, or neuromuscular disorder
2. Thyroid disease
3. History of smoking
4. Alcohol consumption which exceeds 2 drinks per day and /or drug abuse. Volunteers will be asked the question: How many drinks are you drinking on your typical day?
5. Allergy to study medication (propofol), soy, or egg proteins.
6. History of drug abuse
7. Chronic or acute use of opioids, or other medications affecting the CNS
8. Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical efficacy of the ReinLoop agent in delivering closed-loop, patient-specific hypnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Doufas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States